CLINICAL TRIAL: NCT07377318
Title: Methods to Enhance Caregivers' Knowledge of Alzheimer's Disease and Related Dementias (ADRD)
Brief Title: Project CARE-D - Online Caregiver Education for Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Uma Tauber, Professor of Psychology, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-153
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dementia
Keywords: dementia care
MeSH Terms: conditions — Dementia | interventions — Commerce

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants are masked to study hypothesis. Analyses are conducted blind to condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Retrieval Practice (SRP) (Experimental)
  Interventions: Behavioral: Structured Retrieval Practice
- Standard Retrieval Practice (Active Comparator)
  Interventions: Behavioral: Standard Retrieval Practice
- Self-paced Study (Active Comparator)
  Interventions: Behavioral: Business as usual learning

INTERVENTIONS:
Behavioral: Structured Retrieval Practice — The primary learning principle driving the proposed learning intervention is retrieval practice. The efficacy of spaced retrieval practice for learning is supported by a large and robust literature. Accurately recalling information during practice increases the probability that information will be accessible later when the stakes are higher. Caregivers studied all 12 BPSD in the learning phase, at their own pace, and then completed retrieval practice trials by answering multiple choice questions. Each multiple choice question had 1 correct answer and 3 incorrect lures. Detailed, corrective, and elaborative feedback was provided after each response to reinforce correct answers and correct wrong responses. The order of learning strategy was randomized per caregiver, and caregivers went through the learning phase a total of three times. Strategy was consistent between trials.
  Arms: Structured Retrieval Practice (SRP)
Behavioral: Business as usual learning — Caregivers were informed that they would read about 12 BPSD and that they should try their best to read each text as if they were researching the material on their own. Caregivers then studied each of the 12 BPSD, one-by-one, in a webpage format, at their own pace.
  Arms: Self-paced Study
Behavioral: Standard Retrieval Practice — Caregivers completed retrieval practice trials during learning by responding to multiple choice questions each with 1 correct answer and 3 incorrect lures. No feedback was provided following their response selections.
  Arms: Standard Retrieval Practice

SUMMARY:
Managing daily symptoms for people with Alzheimer's Disease or Related Dementia (ADRD) can be challenging and confusing for informal caregivers who are family members or friends and not paid for their assistance. This is due, in part, to gaps in knowledge. Ensuring that informal caregivers are properly educated about ADRD symptoms and treatment guidelines is an essential first step for reducing adverse health events that people living with ADRD experience and addressing the substantial emotional and physical burden that caregivers report. The goal of is project is to improve caregiver education to support treatment adherence for ADRD with retrieval practice. This intervention incorporates principles from the science of learning for structuring retrieval practice to optimize learning and that are effective across the lifespan to compensate for gaps in knowledge and processing capabilities including learners who experience associative memory deficits due to age, their own disease state, or other factors.

ELIGIBILITY:
Inclusion Criteria:

* informal caregivers
* located in the United States
* Speak and read English
* free of cognitive deficits that would prevent consenting and/or completing online experimental tasks

Exclusion Criteria:

* formal caregivers
* former caregivers who are not currently in a care role for a person living with dementia
* technology issues that cause loss of data (e.g., internet connection failure)
* not finishing the experiment
* significant distractions during experimental tasks
* failure to pass attention or bot checks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Delayed test performance | 2 days following first session
  proportion correct on the final 2-day delayed test of symptoms and treatments of ADRD. The test will be in multiple-choice format.
Immediate test performance | at the end of the first session; 10 minutes post-intervention
  proportion correct on the immediate (approx. 10 min retention interval) test of symptoms and treatments of ADRD. The test will be in multiple-choice format.

SECONDARY OUTCOMES:
caregiver self-efficacy | 2 days following intervention (i.e., session 2 measure)
  Caregiver self-efficacy for symptom management will be measured using the symptom subscale of the Family Caregiver Self-efficacy for Dementia Scale, which includes 5 items. An example item is, "how certain are you right now that you can handle any problems your relative has, like memory loss, wandering, or behavior problems." Responses will be given using a 1 (not at all certain) to 10 (very certain) scale. We will expand this scale to include items that match with our content and our symptom presence, severity, and frequency measure. Specifically, participants will respond to 12 questions using a scale from 1 (not at all certain) to 10 (very certain). An example item is, "how certain are you right now that you can handle when your loved one living with dementia experiences false beliefs or delusions?"
E-Health Literacy | 2 days following intervention (i.e., session 2 measure)
  The E-health Literacy Scale (eHEALS) will be administered to assess perceived skills and comfort related to using internet resources for acquiring health knowledge. The scale includes 10 questions (e.g., I can tell high quality from low quality health resources on the internet). Questions require responding on a Likert sale ranging from 1 to 5 (1-strongly disagree, 2- disagree, 3-undecided, 4-agree, 5-strongly agree; 1-not useful at all, 2-not useful, 3-unsure, 4-useful, 5-very useful; or 1-not important at all, 2-not important, 3-unsure, 4-important, 5-very important). Composite scores will be calculated with higher scores indicate higher e-health literacy.
Letter and pattern comparison | 2 days following intervention (i.e., session 2 measure)
  Perceptual speed will be measured with the Letter Comparison Test and Pattern Comparison Test. The Letter Comparison Test involves 21 letter string pairs to be judged as the same or different. The Pattern Comparison Test involves 30 line patterns to be judged as the same or different. For both comparison tests, participants are given 24 seconds per test to complete as many items as possible, and performance is calculated as the number of items correct. Performance on each test will be calculated as the number of items correct, and a composite score will be calculated per participant.
Raven's progressive matrices | immediately following the intervention
  Non-verbal fluid intelligence will be assessed with a computerized version of Raven's progressive matrices. Participants will complete 18 trials in ascending order in trial normative difficulty . For each trial, a 3 x 3 array will be displayed with 8 geometric figures. The 9th position in the bottom right-hand corner will be empty. Participants will be given 8 geometric figures from which to choose to correctly complete the array. Participants will be given 10 minutes to complete as many trials as possible. Performance will be calculated as the total number of trials correct.
Vocabulary | 2 days following intervention (i.e., session 2 measure)
  General knowledge will be assessed using a common measure of general knowledge in cognitive aging research, the Advanced Vocabulary Test I-v-4 . Participants will be presented with a series of words and required to select the synonym for each word out of five options. Participants are given 4 min per task to complete as many words as possible (36 total problems, 8 min total). The self-paced vocabulary test is presented in a fixed order, and no feedback is provided. Performance is calculated as the number of items correct while adjusting for guessing (i.e., number of items correct - (.2 * number of items incorrect)).
Medical health knowledge | 2 days following intervention (i.e., session 2 measure)
  Participants will complete the Medical Term Recognition Test. The METER is completed on paper. A list of 40 medical words and 40 nonwords are presented. Participants read the list of items and select the ones that they recognize as real words. Participants are instructed not to guess and to only select items they are sure were real words. Performance on the METER is calculated as the number of words correctly recognized.
Performance during learning | Baseline
  Caregivers' performance during learning will be defined as the percent correct on retrieval practice trials. Specifically, caregivers will respond to multiple choice questions during learning when engaging in retrieval practice, and learning progress will be quantified by aggregating responses across items for each block. Each multiple choice question will have 1 correct answer and 3 incorrect lures, and responses will be scored as 1 (correct) or 0 (incorrect) and then aggregated per participant. This is a quantitative measure that is standard in the science of learning and for which no validated scale is available. Performance on retrieval practice trials for the will be evaluated with item-level analysis (to explore content difficulty) and across each learning block to establish participants' rate-of-learning.
Symptom presence, severity, and frequency | 2 days following intervention (i.e., session 2 measure)
  The behavioral and psychological symptoms experienced by the person living with dementia will be rated by the caregiver participants using the updated version of the Neuropsychiatric Inventory Questionnaire (NPI-Q). This measure includes 12 items that the participant will rate on presence (yes vs. no), severity (1 = mild, 2 = moderate, 3 = severe), and distress (1 = not distressing at all to 5 = extremely distressing).
Usability measures | Baseline
  The Technology Acceptance Model (TAM) 3 scale will be administered, and scale composite score will be calculated. Example items are, "I find this system easy to use." and "The actual process of using the system is pleasant." Minor adaptations will be implemented to ensure questions are applicable to dementia care. Responses to all questions will be made on a 7-point Likert scale from strongly disagree to strongly agree.
Demographic characteristics | Baseline and 2 days following baseline
  This is not a scale measure, and no composite score or subscores are calculated. Instead, these are descriptive data about the sample so they are accurately described for considerations of generalizability. Questions include: age, gender, education level, race/ethnicity, first generation status, member of an underrepresented group, native language, socioeconomic status, occupation, relationship with individual living with Alzheimer's Disease or a related dementia (e.g., child, spouse), information seeking about dementia and caregiving, and duration of caregiving
self-reported subjective health information | Baseline
  Caregivers will self-report co-morbid medical conditions for the PLwD, and will report medication use, rating of health, hospitalizations, access to health insurance for the PLwD. Caregivers will be allowed to skip any questions they desire should they prefer not to report responses to any of these questions. No measurement scale will be used for these self-report questions. Instead, these brief questions are intended to obtain general health information. Example questions include, "does the person have other chronic conditions?" "Does the person living with dementia take any prescription medications?" and "Have you gone to the hospital emergency room (ER) about the person living with dementia's health in the past year (12 months)?" Responses to these questions will be used for descriptive purposes to better understand the sample and will not be aggregated into one measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Fortinsky, R. H., Kercher, K., & Burant, C. J. (2002). Measurement and correlates of family caregiver self-efficacy for managing dementia. Aging & Mental Health, 6(2), 153-160. doi:10.1080/13607860220126763
- [Background] Venkatesh, V., & Bala, H. (2008). Technology Acceptance Model 3 and a Research Agenda on Interventions. Decision Sciences, 39(2), 273-315. doi: 10.1111/j.1540-5915.2008.00192.x
- [Background] Ariel, R., Babineau, A., & Tauber, S. K. (2023). Teaching older adults to use retrieval practice improves their self-regulated learning. Aging, Neuropsychology, and Cognition, 31(5), 823-845. doi: 10.1080/13825585.2023.2271531
- [Background] Stanovich, K. E., & Cunningham, A. E. (1993). Where does knowledge come from? Specific associations between print exposure and information acquisition. Journal of Educational Psychology, 85(2), 211. doi: 10.1037/0022-0663.85.2.211
- [Background] Kaufer, D.I., Cummings, J.L., Ketchel, P., Smith, V., MacMillan, A., Shelley, T., Lopez, O.L., & DeKosky, S.T. (2000). Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. Journal of Neuropsychiatry and Clinical Neuroscience, 2(2), 233-239. doi: 10.1176/jnp.12.2.233.
- [Background] Salthouse, T. A., & Babcock, R. L. (1991). Decomposing adult age differences in working memory. Developmental Psychology, 27(5), 763-776. doi: 10.1037/0012-1649.27.5.763.
- [Background] Rawson, K. A., Gunstad, J., Hughes, J., Spitznagel, M. B., Potter, V., Waechter, D., Rosneck, J. (2010). The METER: A Brief, self-administered measure of health literacy. Journal of General Internal Medicine, 25, 67-71. doi:10.1007/s11606-009-1158-7
- [Background] Ekstrom, R. B., French, J. W., Harmon, H. H., & Dermen, D. (1976). Manual for kit of factor-referenced cognitive tests. Educational Testing Service.
- [Background] Raven, J., Raven, J. C., & Court, J. H. (1998). Raven manual section 4: Advanced progressive matrices. Oxford. Oxford University Press.
- [Background] Norman, C. D., & Skinner, H. A. (2006). eHEALS: The eHealth literacy scale. Journal of Medical Internet Research, 8(4), e507. doi: 10.2196/jmir.8.4.e27
- [Background] Woods, S. P., Babicz, M. A., Matchanova, A., Sullivan, K. L., Avci, G., Hasbun, R., Giordano, T. P., Fazeli, P., & Morgan, E. E. (2021). A clinical pilot study of spaced retrieval practice with a self-generation booster to improve health-related memory in persons with HIV disease. Archives of Clinical Neuropsychology, 36(7), 1296-1306. doi: 10.1093/arclin/acaa130
- [Background] Tse, C., Balota, D. A., & Roediger, H. L. (2010). The benefits and costs of repeated testing on the learning of face-name pairs in healthy older adults. Psychology and Aging, 25(4), 833-845. doi:10.1037/a0019933
- [Background] Sumowski, J. F., Wood, H. G., Chiaravalloti, N., Wylie, G. R., Lengenfelder, J., & Deluca, J. (2010). Retrieval practice: A simple strategy for improving memory after traumatic brain injury. Journal of the International Neuropsychological Society, 16(6), 1147-1150. doi: 10.1017/S1355617710001128
- [Background] Ringer, T. J., Wong-Pack, M., Miller, P., Patterson, C., Marr, S., Misiaszek, B., Woo, T., Sztramko, R., Vastis, P. G., & Papaioannou, A. (2020). Understanding the educational and support needs of informal caregivers of people with dementia attending an outpatient geriatric assessment clinic. Aging and Society, 40(1), 205-228. doi: 10.1017/S0144686X18000971
- [Background] Jorge, C., Ceto, M., Arias, A., Blasco, E., Gil, M. P., Lopez, R., Dakterzada, F., Purroy, F., & Pinol-Ripoll, G. (2021). Levels of understanding of Alzheimer disease among caregivers and the general population. Neurologia, 36(6), 426-432. doi: 10.1016/j.nrleng.2018.03.004
- [Background] Hernández, M. H., Mestres, C., Modamio, P., Junyent, J., Costa-Tutusaus, L., Lastra, C. F., & Mariño, E. L. (2019). Adverse drug events in patients with dementia and neuropsychiatric/behavioral, and psychological symptoms, a one-year prospective study. International Journal of Environment Research and Public Health, 16(6), 934. doi: 10.3390/ijerph16060934